CLINICAL TRIAL: NCT03820908
Title: Bisantrene for Relapsed /Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Bisantrene for Relapsed /Refractory AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Race Oncology Ltd (Industry)
Responsible Party: Principal Investigator, Prof Arnon Nagler, Arnon Nagler, M.D., M.Sc Professor of Medicine Tel Aviv University, Director Hematology Division BMT and Cord Blood Bank, Chair Israeli BMT Association, Chair of the ALWP of the EBMT, Co-Chair Scientific Council of the EBMT, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5792-18 - SMC
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Acute Myelogenous Leukemia; Allogeneic Stem Cell Transplantation
Keywords: relapsed AML; refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — bisantrene

STUDY DESIGN:
Intervention Model Description: The patientswith Rel /Ref AML will receive bisantrene in conjunction with the conventional supportive care. In the event of a CR, patients will receive a 3-day consolidation course of bisantrene 250mg/m2/d (optional).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bisantrene (Experimental): patients will receive bisantrene 250mg/m2/d for 7 days
  Interventions: Drug: Bisantrene

INTERVENTIONS:
Drug: Bisantrene — The patients will receive bisantrene 250mg/m2/d for 7 days in conjunction with the conventional supportive care.

SUMMARY:
Induction of response in patients with AML that are either primary resistant (failed induction and or salvage therapy) or relapsed including post allogeneic stem cell transplantation and failed salvage therapy or cannot receive additional anthracycline .

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible to enroll in this study.

Disease-related:

1. Patients with Rel/Ref/AML
2. Adequate birth control in fertile patients.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Demographic:

1. Age ≥ 18 years and willing and able to comply with the protocol requirements
2. Life expectancy ≥ 3 months Ethical/Other
3. Written informed consent in accordance with federal, local, and institutional guidelines.
4. Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception.
5. Male subjects must agree to practice contraception

Exclusion Criteria:

* Disease-related

  1. Patients with other type of basic disease other than Rel/Ref AML.
  2. Patients with respiratory failure (DLCO < 30%).
  3. Patients with active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention.
  4. Patients with > grade II liver renal toxicity.
  5. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate
  6. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
  7. Creatinine > 2.0 mg/dl
  8. ECOG-Performance status > 2
  9. CNS disease involvement
  10. Severe pleural effusion and ascites. Concurrent Conditions

  <!-- -->

  1. Pregnant or lactating females
  2. Known human immunodeficiency virus infection
  3. Active hepatitis B or C infection
  4. Non hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
  5. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
  6. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.
  7. Patients with relapse or disease progression >3 months post HSCT are allowed into the study unless they have severe (grade III-IV) GVHD.

Patients with grade III-IV GVHD will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | 24 months
  Overall survival will be calculated from the day of bisantrene administration until death or last follow-up.
Leukemia-free survival | 24 months
  Leukemia-free survival will be calculated from the day of bisantrene administration until relapse, death of any cause, or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel